CLINICAL TRIAL: NCT04074993
Title: Brigatinib in ALK-positive NSCLC Identified Via Blood-based Assays
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: JI-YOUN HAN (Other Government)
Collaborators: Seoul National University Hospital (Other); Severance Hospital (Other); Seoul National University Bundang Hospital (Other)
Responsible Party: Sponsor-Investigator, JI-YOUN HAN, Principle Investigator, National Cancer Center, Korea
Organization: National Cancer Center, Korea (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2019-0212
Record Dates: First submitted 2019-08-25; First posted 2019-08-30 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — brigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brigatinib (Experimental): Subject will be treated with Brigatinib 90mg/day for 1 week and then 180mg/day PO daily. A Cycle will be defined as 28-days. Treatment will be continued until disease progression or unacceptable toxicity.
  Interventions: Drug: Brigatinib

INTERVENTIONS:
Drug: Brigatinib — Subject will be treated with Brigatinib 90mg/day for 1 week and then 180mg/day PO daily. A Cycle will be defined as 28-days. Treatment will be continued until disease progression or unacceptable toxicity.

SUMMARY:
This is single-arm, open-label study design. Patients will receive brigatinib until disease progression, unacceptable toxicity, withdrawal of consent, of death.

DETAILED DESCRIPTION:
Based on the clinical efficacy of ALK inhibitors in ALK+NSCLC, NCCN guidelines recommend ALK molecular testing of lung cancer patients, to select patients for ALK-targeted therapy. However, molecular testing via tissue biopsy cannot always be performed on NSCLC patients, potentially limiting access of effective treatment to the subset of patients who are able to undergo current testing procedures that utilize tissue biopsies. Obtaining an adequate tissue biopsy specimen for NSCLC presents a number of challenges. In particular, the method for diagnosis of lung cancer depends on the location, size, and type of suspected lung cancer, and the presence or absence of metastases. Common procedures for centrally located tumors include bronchoscopy and sputum cytology, which frequently yield insufficient tumor tissue for comprehensive mutation testing. In addition, 75% of patients are diagnosed with late-stage disease and often present with multiple comorbidities. Biopsies in these patients can lead to complications such as pneumothorax, hemoptysis, other bleeding complications, and cardiopulmonary decompensation. As a result of these factors, a physician treating a patient who presents with a significant burden of disease as well as significant comorbidities may rightly consider whether it is in the best interest of the patient to undergo a risky and potentially unsuccessful procedure. Thus, there exists a major unmet clinical need for testing procedures that do not require tumor tissue. The purpose of this phase II study is to assess the efficacy of brigatinib in patients with advanced NSCLC harboring ALK rearrangement that are selected using predictive biomarkers identified via blood-based assays.

ELIGIBILITY:
Inclusion Criteria:

1. The participant(or legally acceptable representative if applicable) provides written informed consent for the study
2. Patients who have disease progression with prior one ALK-TKI treatment for inoperable Stage III (locally advanced) or metastatic ALK+ NSCLC.(Previous treatment only allowed one ALK-inhibitor) Patients who have received prior neo-adjuvant, adjuvant chemotherapy, radiotherapy, or chemoradiotherapy with curative intent for non-metastatic disease must have experienced a treatment-free interval of at least 6 months since the last chemotherapy, radiotherapy, or chemoradiotherapy cycle.
3. ALK rearrangement , as detected via the blood somatic mutation assay
4. One prior ALK inhibitor therapy
5. Have at least 1 measurable lesion per RECIST version 1.1
6. Have Eastern Cooperative Oncology Group (ECOG) performance status 0-2
7. Recovered from toxicities related to prior anticancer therapy to NCI CTCAE, version 5.0, Grade≤1(Note : Alopecia, sensory neuropathy Grade≤2, or other Grade≤2 AEs not constituting a safety risk based on Investigator's judgement are acceptable
8. Have a life expectancy of ≥3 months
9. Have adequate organ and hematologic function as determined by:

   1. ALT/AST≤2.5×ULN; ≤5×ULN is acceptable if liver metastases are present
   2. Total serum bilirubin≤1.5×ULN (<3.0×ULN for patients with Gilbert syndrome)
   3. Estimated glomerular filtration rate (eGFR) ≥30 mL/min/1.73 m2, using the MDRD equation
   4. Absolute neutrophil count ≥1.5×109/L.
   5. Platelet count ≥75×109/L.
   6. Hemoglobin ≥9 g/dL.
   7. Serum lipase ≤1.5×ULN
10. For female patients of childbearing potential, have a negative pregnancy test(urine or serum) documented ≤3 days before start of study medication.

    non-childbearing potential which is defined as :
    * female patient≥45 years of age and has not had menses for greater than 1 year
    * a female who is status post hysterectomy, oophorectomy
11. Female patients of childbearing potential and male patients with partners of childbearing potential must agree to use 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 4 months after the last dose of study drug, or agree to completely abstain from heterosexual intercourseHave the willingness and ability to comply with scheduled visit and study procedures.

    Male patients, even if surgically sterilized (i.e., status post-vasectomy), who:
    * Agree to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug, or
    * Agree to completely abstain from heterosexual intercourse
12. Have the willingness and ability to comply with scheduled visit and study procedures.
13. Be ≥ 18 years of age

Exclusion Criteria:

1. Has received ALK-targeted TKI within 7 days before the first dose of study treatment(If clinically justified, 3 days wash-out period could be allowed).
2. Has received radiotherapy within 14 days before the first dose of study treatment except for stereotactic radiosurgery (SRS) or stereotactic body radiation therapy (SBRT). A 1-week washout is permitted for palliative radiation(≤2 weeks of radiotherapy) to non-CNS disease.
3. Had major surgery within 28 days of the first dose of study treatment. Minor surgical procedures are allowed.
4. Has symptomatic brain metastasis or leptomeningeal disease. Prior brain metastasis or leptomeningeal disease allowed if asymptomatic or stable symptoms that did not require an increased dose of corticosteroids to control symptoms within 7 days prior to study enrollment. If patients have neurological symptoms or signs due to CNS metastasis, patients need to complete whole brain radiation or stereotactic radiosurgery treatment before enrollment and be clinically stable.
5. Has current spinal cord compression
6. Other malignancy within 3 years, except for adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, and ductal carcinoma in situ treated surgically with curative intent
7. Any gastrointestinal (GI) disorder that may affect absorption of oral medications, such as malabsorption syndrome or status post-major bowel resection
8. Have significant, uncontrolled, or active cardiovascular disease, specifically including, but not restricted to:

   1. Myocardial infarction within 6 months before the first dose of brigatinib.
   2. Unstable angina within 6 months before first dose of brigatinib.
   3. Congestive heart failure within 6 months before first dose of brigatinib.
   4. History of clinically significant atrial arrhythmia (including clinically significant bradyarrhythmia).
   5. Any history of clinically significant ventricular arrhythmia.
9. Has uncontrolled hypertension.
10. Had a cerebrovascular accident or transient ischemic attack within 6 months before first dose brigatinib.
11. Have a history or the presence of pulmonary interstitial disease, drug-related pneumonitis, or radiation-related pneumonitis
12. Active infection requiring systemic therapy.
13. Known history of HIV infection.
14. Has a known or suspected hypersensitivity to brigatinib or its excipients.
15. Female patients who are both lactating and breastfeeding or have a positive serum pregnancy test during the screening period or a positive urine pregnancy test on Day 1 before first dose of study drug (if applicable).
16. Have any condition or illness that, in the opinion of the investigator, would compromise
17. patient safety or interfere with the evaluation of brigatinib
18. Received systemic treatment with strong cytochrome P-450 (CYP)3A inhibitors, strong CYP3A inducers, or moderate CYP3A inducers within 14 days before enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-05-15 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | From Cycle1 Day 1 until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months. Tumor assessment will be performed at the end of cycle 2(every 2 cycles, each cycle is 28 days).
  Objective response rate

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No